CLINICAL TRIAL: NCT06250231
Title: Knowledge and Attitude Towards Fertility Among Emirati Infertile Patients
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2308-ABU-016-AS
Record Dates: First submitted 2023-12-06; First posted 2024-02-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female; Infertility, Male
Keywords: surveys and questionnaires
MeSH Terms: conditions — Infertility, Female; Infertility, Male

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Infertility is on the rise worldwide due to multiple reasons. Proper and timely diagnosis makes the treatment easier and more acceptable by the couple. Lack of fertility knowledge however delays necessary investigations and sometimes reduces chances of success as a consequence of a delay in patients / couples approaching infertility clinics. Assessing the fertility knowledge of the Emirati infertility patients would help us to understand better the cultural aspects of fertility, the driving forces for having children and how much patients actually know about predisposing factors for infertility. This in turn would improve counseling and possible set knowledge campaigns to increase awareness.

ELIGIBILITY:
Inclusion Criteria:

* United Arab Emirates nationals coming for their first consultation in ART Fertility Clinics
* Any age group
* males and females

Exclusion Criteria:

- none

Kindly note that ART is the name of the fertility clinic and not an abbreviation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is the infertile patients seeking In- Vitro Fertilization (IVF) treatment in ART fertility clinics in Abu Dhabi
  Kindly note that ART is the name of the fertility clinic and not an abbreviation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Understanding Knowledge and Attitudes of Emirati Infertility Patients Towards Fertility Issues | 1 year
  A self-built survey was created to cover the different aspects of United Arab Emirates culture. The survey was pilot tested on 9 people not related to the fertility clinic for comprehension and ease of reading. The nature of the questions included would help in understanding the way the local population thinks about fertility in general given that the Emirati society is governed by certain religious and social norms and expectations. The data that will be collected by the end of this study will aid in creating certain guidelines easing the approach to infertile patients as well raising fertility awareness campaigns to encourage patients seek fertility specialist opinion early on that could potentially improve the success rates of fertility treatments.

CONTACTS AND LOCATIONS:
Locations (2):
- United Arab Emirates (2):
  - ART Fertility Clinics, Abu Dhabi
  - ART Fertility Clinics Al Ain, Al Ain City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haynes, D. (2016). ScholarWorks Delaying First Pregnancies: Canadian Women' s Knowledge and Perception of the Consequences. https://scholarworks.waldenu.edu/dissertations
- [Result] Cramer DW, Walker AM, Schiff I. Statistical methods in evaluating the outcome of infertility therapy. Fertil Steril. 1979 Jul;32(1):80-6. PMID 456633
- [Result] Richardson SJ, Senikas V, Nelson JF. Follicular depletion during the menopausal transition: evidence for accelerated loss and ultimate exhaustion. J Clin Endocrinol Metab. 1987 Dec;65(6):1231-7. doi: 10.1210/jcem-65-6-1231. PMID 3119654
- [Result] Rangel EL, Castillo-Angeles M, Easter SR, Atkinson RB, Gosain A, Hu YY, Cooper Z, Dey T, Kim E. Incidence of Infertility and Pregnancy Complications in US Female Surgeons. JAMA Surg. 2021 Oct 1;156(10):905-915. doi: 10.1001/jamasurg.2021.3301. PMID 34319353
- [Result] Blair I, Sharif AA. Population structure and the burden of disease in the United Arab Emirates. J Epidemiol Glob Health. 2012 Jun;2(2):61-71. doi: 10.1016/j.jegh.2012.04.002. Epub 2012 May 22. PMID 23856422
- [Result] Melado L, Vitorino R, Coughlan C, Bixio LD, Arnanz A, Elkhatib I, De Munck N, Fatemi HM, Lawrenz B. Ethnic and Sociocultural Differences in Ovarian Reserve: Age-Specific Anti-Mullerian Hormone Values and Antral Follicle Count for Women of the Arabian Peninsula. Front Endocrinol (Lausanne). 2021 Oct 21;12:735116. doi: 10.3389/fendo.2021.735116. eCollection 2021. PMID 34745004
- [Result] Green KE, Smith DE. Change and continuity: childbirth and parenting across three generations of women in the United Arab Emirates. Child Care Health Dev. 2007 May;33(3):266-74. doi: 10.1111/j.1365-2214.2006.00667.x. PMID 17439440